CLINICAL TRIAL: NCT07092761
Title: Evaluation of the Accuracy and Safety of A Novel Real-Time Continuous Glucose Monitoring System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Peng Liu, Physician, The First Affiliated Hospital of Henan University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SS-KY-CGM-0003
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients with T1DM or T2DM (Other)
  Interventions: Device: GS3 CGM

INTERVENTIONS:
Device: GS3 CGM — Wearing CGM for a consecutive 14 days

SUMMARY:
The study is to evaluate the accuracy and safety of a novel real-time CGM system among adult patients with type 1 diabetes mellitus with respect to YSI reference venous plasma sample measurements.

DETAILED DESCRIPTION:
The study is to evaluate the accuracy and safety of a novel real-time CGM system among adult patients with type 1 diabetes mellitus with respect to YSI reference venous plasma sample measurements. Up to 42 patients will be enrolled. Each patient will wear two sensors. Interstitial glucose readings from each sensor will be obtained immediatedly following each venous blood sample test. Each participant will make 4 visits to the clinical study site, including the screening visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagonsed with T1DM or T2DM
* Venous blood sampling access can be established in the forearm
* Capable of independently reading instructions and complying with the clinical trial requirements
* Willing to sign the Informed Consent Form (ICF)

Exclusion Criteria:

* Severe hypoglycemia within the past 6 month
* Heart failure or hemiplegic sequelae due to prior cerebrovascular disease
* Severe skin conditions at the sensor wear site
* Extensive systemic skin disorders
* Coagulation disorders confirmed by the investigator
* Anemia or abnormal hematocrit
* Blood donation within the past 6 months
* Pregnancy (defined as positive urine test in women ≤55 years), lactation, or plans for pregnancy within ≤30 days
* Current or recent (≤1 month) participation in other clinical trials
* Planned MRI/CT scans during sensor wear
* Allergy to medical adhesives or alcohol
* Conditions impairing comprehension of informed consent or study procedures
* Other exclusionary conditions per investigator's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
System performance | 14 days
  The CGM system performance will be assessed by comparing to the Yellow Springs Instrument comparator venous plasma measurements
System-related Safety | 14 days
  The CGM system will be characterized by adverse device effects experienced by the study participants

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Jiang, Principal Investigator — Henan University of Science and Technology
Locations (1):
- Henan University of Science and Technology, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: No